CLINICAL TRIAL: NCT00534872
Title: A Single-centre, Open Label, Single-dose, Four Parallel Cohorts Study to Investigate the Pharmacokinetics, Safety and Tolerability of SB-649868 10mg in Healthy Female "Non-childbearing Potential", Healthy Male and in Healthy Elderly Subjects
Brief Title: A Clinical Study to Evaluate the Pharmacokinetic Profile of SB-649868 in Elderly and Female Population
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stoppend before recruitment start for preclinical safety finding in rats.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXS109143
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Insomnia
Keywords: 4 Parallel cohorts; Healthy Female; Healthy Elderly; Pharmacokinetic; Safety and Tolerability
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — N-((1-((5-(4-fluorophenyl)-2-methyl-4-thiazolyl)carbonyl)-2-piperidinyl)methyl)-4-benzofurancarboxamide

ARMS (1):
- SB649868 (Experimental): 10 mg
  Interventions: Drug: SB-649868

INTERVENTIONS:
Drug: SB-649868 — 10 mg

SUMMARY:
The purpose of this study is to determine the blood levels and the tolerability of SB-649868 in Elderly and Female population

ELIGIBILITY:
INCLUSION CRITERIA:

* Healthy adult and elderly female and male
* Female must be of non-childbearing potential
* Body weight =50 kg

EXCLUSION CRITERIA:

* Abuse of alcohol or drugs
* Positive for Hepatitis B surface antigen, Hepatitis C antibody or HIV
* Use of prescription or non-prescription drugs within 7 days prior to the first dose of study medication
* Smoking history of = 10 cigarettes a day in the last three months
* History of cardiovascular,psychiatric,autoimmune, respiratory or relevant gastrointestinal diseases
* Participation in clinical trial during the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2007-10 (Estimated); Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Blood levels after a single dose of SB-649868 after 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours | single dose of SB-649868 after 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours

SECONDARY OUTCOMES:
Adverse Event, laboratory, vital signs and ECG abnormality occurred within 7-14 days from a single dose of SB-649868 | within 7-14 days from a single dose of SB-649868

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline